CLINICAL TRIAL: NCT01524042
Title: Patient Satisfaction With Novel Double Pants Compared to Conventional Single Pants for Outpatient Colonoscopy: Prospective Randomized Study
Brief Title: Patient Satisfaction With Novel Double Pants Compared to Conventional Single Pants for Outpatient Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 4-2011-0644
Record Dates: First submitted 2012-01-24; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Colonoscopy
Keywords: Satisfaction; colonoscopy; double pants; single pants
MeSH Terms: conditions — Personal Satisfaction | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- group 2 (Experimental): study group:double pants group
  Interventions: Procedure: Pants for colonoscopy

INTERVENTIONS:
Procedure: Pants for colonoscopy — We divide the patients into group 1 and group 2. The group 1 wear a conventional single pants and group 2 wear a novel double pants.

SUMMARY:
Recently colonoscopy has gained importance as screening programs for colon polyp, cancer and inflammatory bowel disease in the United States and other countries. The number of colonoscopy performed has been increased year by year. To make an increased compliance with colonoscopy in both screening and clinical surveillance programs, consideration of anxiety, shame and satisfaction in examinee is regarded to be important. During colonoscopy patients wear conventional single pants where there is no hole for insertion of scope. Patients take off the conventional single pants below the buttocks and expose their buttocks and perianal area during colonoscopy. Exposing perianal and perineal area during colonoscopy can make patients feel shameful and anxious and diminish satisfaction of colonoscopy. Recently considering the factors affecting satisfaction has been regarded to be important because patient satisfaction could be one of the quality indicators for colonoscopy. To diminish shame and anxiety by exposing perianal and perineal area of patients wearing conventional single pants during colonoscopy, we developed novel double pants with a hole in inner pants. Novel double pants are composed of double fabrics from hip to thigh and single fabric under the thigh such as common pants. In the inner pants of double pants, there is a hole for insertion of scope. The hole is 25 cm wide and 15 cm long. The outer pants are same as conventional single pants. If the patients dropped outer pants below hips, only hip and perianal area are exposed through the hole (25cm*15 cm) for insertion of scope without dropping inner pants. Therefore novel double pants minimized the exposed area of hips than conventional single pants because hips are exposed only the hole of inner pants. Smaller exposed area of hips by novel double pants can minimized the shame and anxiety by diminishing exposing perianal and perineal area during colonoscopy. Therefore advantage of novel double pants is decreasing shame and anxiety and increasing satisfaction by minimizing the exposed area of perianal and perineal area compared with conventional single pants. This study is a randomized controlled study. The investigators will survey the examinees older than 20 years who performed the colonoscopy at Severance Hospital from Feb. 2012 to Jul. 2012 to compare the effect on the satisfaction, shame, and anxiety during colonoscopy between the two groups.

DETAILED DESCRIPTION:
Eighty examinees will wear conventional single pants and another eighty examinees will wear novel double pants randomly. Examinees who underwent colonoscopy within 3 years, with history of bowel resection surgery, cancer, colostomy or ileostomy, psychotic disease such as depression, anxiety disorder, obsessive disorder, treated with emergent colonoscopic procedure, and pregnant or lactating women, an illiterate person and foreigners will be excluded. Questionnaires before colonoscopy are educational background, martial status, indication of colonoscopy, examinee's preference of doctor's gender, and State-trait anxiety level of examinee. Questionnaires after colonoscopy are shame and trait anxiety level, and satisfaction of examinee during colonoscopy. We will also investigate colonoscopy specific quality Indicators such as the ASA status (American society of anesthesiologist's physical status), complications, procedure success. Finally we will compare the difference of satisfaction, shame, and anxiety during colonoscopy between examinees wearing novel double pants and conventional single pants

ELIGIBILITY:
Inclusion Criteria:

* patients older than 20 years who performed colonoscopy at Severance hospital

Exclusion Criteria:

* patients who underwent colonoscopy within 3 years
* patients with Psychotic problems
* patients with colostomy or ileostomy
* patients with bowel resection
* patients who needed emergent colonoscopy
* pregnant women
* lactating women
* illiterate person
* foreigners

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Satisfaction of patients during colonoscopy | 10 minutes after colonoscopy
  We measure the satisfaction during colonoscopy by questionnares

SECONDARY OUTCOMES:
shame and anxiety of patient during colonoscopy | 20 minutes after colonoscopy
  We measure the satisfaction during colonoscopy by questionnares

CONTACTS AND LOCATIONS:
Overall Officials: Soo Jung Park, Dr., Study Director — Severance Hospital
Locations (1):
- Soo Jung Park, Seoul, South Korea